CLINICAL TRIAL: NCT03585764
Title: Phase I Clinical Trial of Adoptive Transfer of Autologous Folate Receptor - Alpha Redirected T Cells for Recurrent High Grade Serous Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: MOv19-BBz CAR T Cells in aFR Expressing Recurrent High Grade Serous Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was halted prematurely due to recruitment barriers
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH); OvaCure Fundation (Unknown); Alliance for Cancer Gene Therapy (Other); Ovarian Cancer Alliance of Greater Cincinnati (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 830111 (UPCC-03818); 1R01CA260902 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Cohort 1: MOv19-BBz CAR T cells without chemo (Experimental): Cohort 1: (n= 3 to 6 subjects): Single infusion of 1-3x107 /m2 lentivirally transduced MOv19-BBz CAR T cells on day 0 without lymphodepleting chemotherapy.
  Interventions: Drug: MOv19-BBz CAR T cells; Device: Alpha Folate Receptor expression test
- Cohort 2: MOv19-BBz CAR T cells after chemo (Experimental): Cohort 2: (n= 3 to 6 subjects): Single infusion of 1-3x107 /m2 lentivirally transduced MOv19-BBz CAR T cells on day 0 beginning 3 days (+/- 1 day) after lymphodepleting chemotherapy with cyclophosphamide + fludarabine.
  Interventions: Drug: MOv19-BBz CAR T cells; Device: Alpha Folate Receptor expression test
- Cohort 3: MOv19-BBz CAR T cells after chemo (Experimental): Cohort 3: (n=3 to 6 subjects): Single infusion of 1-3x108 lentivirally transduced MOv19-BBz CAR T cells on day 0 beginning 3 days (+/- 1 day) after lymphodepleting chemotherapy with cyclophosphamide + fludarabine.
  Interventions: Drug: MOv19-BBz CAR T cells; Device: Alpha Folate Receptor expression test
- Cohort-1: without chemo;only if dose de-escalation required (Experimental): Cohort -1: (n= 3 to 6 subjects): Single Infusion of 1-3x106 /m2 lentivirally transduced MOv19-BBz CAR T cells on day 0 without lymphodepleting chemotherapy. Up to 6 subjects will be infused in Cohort -1 with ≤ 1 DLT/6 subjects to establish the MTD.
  Interventions: Drug: MOv19-BBz CAR T cells; Device: Alpha Folate Receptor expression test

INTERVENTIONS:
Drug: MOv19-BBz CAR T cells — intraperitoneally administered lentiviral transduced MOv19-BBz CAR T cells with or without cyclophosphamide + fludarabine as lymphodepleting chemotherapy.
Device: Alpha Folate Receptor expression test — Patients will first be pre-screened for alpha folate receptor expression. The test for alpha folate receptor expression is a laboratory developed test+, developed and conducted by the Hospital of the University of Pennsylvania Pathology and Laboratory Medicine lab to determine subject eligibility. This test is not an approved FDA device and its use is investigational.

SUMMARY:
Phase I study to establish safety and feasibility of intraperitoneally administered lentiviral transduced MOv19-BBz CAR T cells with or without cyclophosphamide + fludarabine as lymphodepleting chemotherapy

DETAILED DESCRIPTION:
This is a Phase I study evaluating the safety and feasibility of intraperitoneally administered lentiviral transduced MOv19-BBz CAR T cells in 4 cohorts with or without cyclophosphamide + fludarabine in a 3+3 dose escalation design.

The DLT observation period is 28 days post CAR T cell infusion. The Maximum Tolerated Dose (MTD) is defined as the dose at which 0 or 1 DLT occurs in 6 evaluable subjects tested within the dose range of this study.

Cohort 1: (n= 3 to 6 subjects): Single infusion of 1-3x107 /m2 lentivirally transduced MOv19-BBz CAR T cells on day 0 without lymphodepleting chemotherapy.

Cohort 2: (n= 3 to 6 subjects): Single infusion of 1-3x107 /m2 lentivirally transduced MOv19-BBz CAR T cells on day 0 beginning 3 days (+/- 1 day) after lymphodepleting chemotherapy with cyclophosphamide + fludarabine.

Cohort 3: (n=3 to 6 subjects): Single infusion of 1-3x108 lentivirally transduced MOv19-BBz CAR T cells on day 0 beginning 3 days (+/- 1 day) after lymphodepleting chemotherapy with cyclophosphamide + fludarabine.

Cohort -1: (n= 3 to 6 subjects): Single Infusion of 1-3x106 /m2 lentivirally transduced MOv19-BBz CAR T cells on day 0 without lymphodepleting chemotherapy. Up to 6 subjects will be infused in Cohort -1 with ≤ 1 DLT/6 subjects to establish the MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed persistent or recurrent stage II to IV high grade serous epithelial ovarian, fallopian tube or primary peritoneal carcinoma. Disease can be platinum-sensitive or platinum-resistant.
2. Failure of at least two prior chemotherapy regimens for advanced stage disease. Prior therapies against PD-1 or PDL-1 are permissible.
3. Confirmation of tumor aFR expression (≥70% of tumor cells with ≥2+ aFR staining).
4. Subjects must have measureable disease as defined by RECIST 1.1 criteria.
5. Patients with asymptomatic CNS metastases that have been treated and are off steroids are allowed. They must meet the following at the time of eligibility confirmation by physician-investigator:

   1. No concurrent treatment for the CNS disease
   2. No progression of CNS metastasis on brain MRI at screening
   3. No evidence of leptomeningeal disease or cord compression
6. Patients ≥ 18 years of age.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Satisfactory organ and bone marrow function as defined by the following:

   i. Absolute neutrophil count ≥ 1,000/μl ii. Platelets ≥75,000/μl iii. Hemoglobin ≥ 9 g/dL iv. Total bilirubin ≤ 2.0x the institutional normal upper limit unless secondary to bile duct obstruction by tumor v. Creatinine ≤ 1.5x the institutional normal upper limit vi. Albumin ≥2 vii. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5x the institutional normal upper limit viii. Cardiac ejection fraction of ≥40%
9. Blood coagulation parameters: PT such that international normalized ratio (INR) is ≤ 1.5 and a PTT ≤ 1.2 time the upper limit of normal unless the patient is therapeutically anti-coagulated for history of cancer-related thrombosis and has stable coagulation parameters.
10. Provides written informed consent.
11. Subjects of reproductive potential must agree to use acceptable birth control methods, as described in protocol Section 4.3.

Exclusion Criteria:

1. High grade serous ovarian, fallopian, or primary peritoneal cancer that is platinum refractory, defined as disease that has clinical or radiographic progression on platinum-based chemotherapy, as per the discretion of the treating physician.
2. Patients with symptomatic CNS metastases are excluded.
3. Participation in a therapeutic investigational study within 4 weeks prior to eligibility confirmation by physician-investigator, or anticipated treatment with another investigational product while on study. This refers to non-commercially approved investigational drugs different than those used in this protocol.
4. Active invasive cancer other than ovarian cancers. Patients with active non-invasive cancers (such as non-melanoma skin cancer, superficial cervical and bladder cancer) are not excluded.
5. HIV infection
6. Hepatitis B or hepatitis C infection
7. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to >/= 10 mg of prednisone. Patients with autoimmune neurologic diseases (such as multiple sclerosis) will be excluded.
8. Patients with active and uncontrolled infection.
9. Planned concurrent treatment with systemic high dose corticosteroids. Patients may be on a stable low dose of steroids (<10 mg daily equivalent of prednisone). Corticosteroids treatment as anti-emetic prophylaxis on the day of lymphodepleting chemotherapy administration is allowed per institutional guidance. The use of topical and/or inhaled steroids are not exclusionary.
10. Patients requiring supplemental oxygen therapy.
11. Prior therapy with lentiviral gene modified cells.
12. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
13. Any ascites requiring therapeutic drainage within 4 weeks prior to eligibility confirmation by physician-investigator.
14. Pregnant or breastfeeding women.
15. Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results, and, in the opinion of the physician-investigator, would make the patient inappropriate for entry into the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Payal D Shah, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 Subjects were screen failure and were not assigned to a cohort.
Period: Overall Study
Arm/Group | Cohort 1: MOv19-BBz CAR T Cells Without Chemo | Cohort 2: MOv19-BBz CAR T Cells After Chemo | Cohort 3: MOv19-BBz CAR T Cells After Chemo | Cohort-1: Without Chemo;Only if Dose De-escalation Required
Started | 3 | 3 | 5 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 5 | 0
Not completed — Death | 3 | 2 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Cohort -1 was never opened
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: MOv19-BBz CAR T Cells Without Chemo | Cohort 2: MOv19-BBz CAR T Cells After Chemo | Cohort 3: MOv19-BBz CAR T Cells After Chemo | Cohort-1: Without Chemo;Only if Dose De-escalation Required | Total
Number analyzed (Participants) | 3 | 3 | 5 | 0 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 4 | 0 | 7
  >=65 years | 2 | 1 | 1 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 0 | 11
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 5 | 0 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 5 |  | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Subjects With Treatment-related Adverse Events Using NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Description: For this study, collection of adverse events will begin at the time of apheresis and will continue until the subject is off-study.
Time Frame: Up to 34 months
Population: No participants were enrolled in cohort 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MOv19-BBz CAR T Cells Without Chemo | Cohort 2: MOv19-BBz CAR T Cells After Chemo | Cohort 3: MOv19-BBz CAR T Cells After Chemo | Cohort-1: Without Chemo;Only if Dose De-escalation Required
Number analyzed (Participants) | 3 | 3 | 3 | 0
Participants | 3 | 3 | 3 | 0

2. Primary Outcome: Manufacturing Feasibility
Description: Manufacturing feasibility is determined based on the "manufacturing failures" products. The number of manufactured products that do not meet release criteria for vector transduction efficiency, CART+ cell number, T cell purity, viability, and sterility will be determined and defined as "manufacturing failures".
Time Frame: 8 weeks
Population: No participants were enrolled in cohort -1
Measure: Number; unit: Product manufacture failures
Arm/Group | Cohort 1: MOv19-BBz CAR T Cells Without Chemo | Cohort 2: MOv19-BBz CAR T Cells After Chemo | Cohort 3: MOv19-BBz CAR T Cells After Chemo | Cohort-1: Without Chemo;Only if Dose De-escalation Required
Number analyzed (Participants) | 3 | 3 | 5 | 0
Product manufacture failures | 0 | 0 | 0 |

3. Primary Outcome: Clinical Feasibility
Description: Clinical feasibility is defined as the proportion of subjects enrolled on this protocol who do not receive MOv19-BBz CAR T cells. Reasons for this occurrence include rapid clinical deterioration or death, and subject withdrawal.
Time Frame: 8 weeks
Population: No participants were enrolled in cohort -1. Thirty five (35) participants were enrolled in the study but they screen failed and did not receive MOv19-BBz CAR T cell.
Measure: Number; unit: Participants who didn't receive CART cel
Arm/Group | Cohort 1: MOv19-BBz CAR T Cells Without Chemo | Cohort 2: MOv19-BBz CAR T Cells After Chemo | Cohort 3: MOv19-BBz CAR T Cells After Chemo | Cohort-1: Without Chemo;Only if Dose De-escalation Required
Number analyzed (Participants) | 3 | 3 | 5 | 0
Participants who didn't receive CART cel | 0 | 0 | 2 |

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS will be evaluated up to 5 years post-infusion or until subjects initiate a cancer-related therapy
Time Frame: Up to 33 months
Population: No participants were enrolled in Cohort -1
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 1: MOv19-BBz CAR T Cells Without Chemo | Cohort 2: MOv19-BBz CAR T Cells After Chemo | Cohort 3: MOv19-BBz CAR T Cells After Chemo | Cohort-1: Without Chemo;Only if Dose De-escalation Required
Number analyzed (Participants) | 3 | 3 | 3 | 0
Days | 42 [28 to 86] | 80 [74 to 177] | 21 [18 to 64] |

5. Secondary Outcome: Overall Response Rates (ORR)
Description: ORR is the proportion of subjects with a best response of CR or PR based on RECIST 1.1, as compared to baseline. ORR will be evaluated up to 5 years post-infusion or until subjects initiate a cancer-related therapy.
Time Frame: Up to 33 months
Population: No participants were enrolled in Cohort -1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MOv19-BBz CAR T Cells Without Chemo | Cohort 2: MOv19-BBz CAR T Cells After Chemo | Cohort 3: MOv19-BBz CAR T Cells After Chemo | Cohort-1: Without Chemo;Only if Dose De-escalation Required
Number analyzed (Participants) | 3 | 3 | 3 | 0
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of the infusion to the date of death due to any reason. OS will be evaluated up to 15 years post-infusion.
Time Frame: Up to 33 months
Population: No participants were enrolled in Cohort -1
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 1: MOv19-BBz CAR T Cells Without Chemo | Cohort 2: MOv19-BBz CAR T Cells After Chemo | Cohort 3: MOv19-BBz CAR T Cells After Chemo | Cohort-1: Without Chemo;Only if Dose De-escalation Required
Number analyzed (Participants) | 3 | 3 | 3 | 0
Days | 187 [184 to 248] | 163 [85 to 975] | 136 [18 to 332] |

ADVERSE EVENTS:
Time Frame: Up to 34 months
Description: For this study, collection of adverse events will begin at the time of apheresis and will continue until the subject is off-study. For subjects who do not undergo apheresis on this study (i.e. historical apheresis product available), adverse event reporting period will begin at the time of CAR T cell infusion (Cohorts 1 and -1) or at the start of lymphodepleting chemotherapy (Cohorts 2 and 3). Collection of adverse events will continue until the subject is off-study.
Arm/Group | Cohort 1: MOv19-BBz CAR T Cells Without Chemo | Cohort 2: MOv19-BBz CAR T Cells After Chemo | Cohort 3: MOv19-BBz CAR T Cells After Chemo | Cohort-1: Without Chemo;Only if Dose De-escalation Required
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 3/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 4/5 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MOv19-BBz CAR T Cells Without Chemo (N=3) | Cohort 2: MOv19-BBz CAR T Cells After Chemo (N=3) | Cohort 3: MOv19-BBz CAR T Cells After Chemo (N=5) | Cohort-1: Without Chemo;Only if Dose De-escalation Required (N=0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Acute myeloid leukemia) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MOv19-BBz CAR T Cells Without Chemo (N=3) | Cohort 2: MOv19-BBz CAR T Cells After Chemo (N=3) | Cohort 3: MOv19-BBz CAR T Cells After Chemo (N=5) | Cohort-1: Without Chemo;Only if Dose De-escalation Required (N=0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other (Catheter site pain) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other (Citrate reaction) (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (4) | 4 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 3 (3) | 3 (7) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 3 (4) | 4 (7) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (4) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Morbilliform eruption) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 1 (3) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT03585764/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT03585764/ICF_000.pdf